CLINICAL TRIAL: NCT01838824
Title: Applying Speed of Processing Training (SPT) to Individuals With Multiple Sclerosis
Brief Title: Applying Speed of Processing Training to Individuals With Multiple Sclerosis
Acronym: SPTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Neuropsychology & Neuroscience Lab, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RG 4607-A-3
Record Dates: First submitted 2012-05-11; First posted 2013-04-24 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
Keywords: Processing Speed; Intervention; Multiple Sclerosis; Cognition
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Speed of Processing Training - Group 1 (Experimental): Group 1 will receive speed of processing training immediately following baseline testing. They will have an evaluation immediately following treatment and a long-term follow-up 6 weeks after finishing treatment.
  Interventions: Behavioral: Speed of Processing Training
- Speed of Processing Training - Group 2 (Experimental): Group 2 will receive speed of processing training 6 weeks following baseline testing. They will have an evaluation immediately following treatment and a long-term follow-up 6 weeks after finishing treatment.
  Interventions: Behavioral: Speed of Processing Training

INTERVENTIONS:
Behavioral: Speed of Processing Training — SPT involves trainer-guided practice of computer-based exercises, including Target Detection (indicating presence or absence of targets, identifying targets, etc.) and Discrimination and Localization (performing same/ different discriminations of targets presented very quickly and followed by a masking pattern) 10, 19, 84. Display speed, ranging from 17 to 500 ms, is the primary manipulation during training, which increases task demands and thus demands on PS itself.

SUMMARY:
This pilot study will document the efficacy of a behavioral intervention for Processing Speed (PS) in Multiple Sclerosis (MS), Speed of Processing Training (SPT), which has been successful used in the aging population in several studies. This study will (1) apply a treatment protocol for PS impairments, well-validated in aging, to persons with MS with impaired PS, and document its efficacy on standard neuropsychological (NP) tests (2) assess the effectiveness of the intervention utilizing global measures of daily life, including an objective measure (TIADL) (3) examine the long term impact of SPT. This study is unique in that it will be the first to evaluate the efficacy of a highly-manualized structured behavioral treatment for processing speed deficits in persons with MS utilizing the optimal methodology for carrying out such studies, a randomized clinical trial. Given the prevalence of PS deficits in the MS population and the significant impact such deficits have on everyday functioning, public safety, and overall quality of life, the identification of an effective intervention for PS deficits in MS could have a profound impact on the population and society as a whole.

ELIGIBILITY:
Inclusions:

* diagnosis of Multiple Sclerosis
* fluent in English
* processing speed impairment (based on evaluation).

Exclusions:

* currently taking steroids and /or benzodiazepines
* prior stroke or neurological disease
* history of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder, Schizophrenia, Bipolar Disorder I or II
* significant alcohol or drug abuse history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-11; Primary Completion 2020-03 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Change in scores on standardized tests of processing speed | Three points in time: Baseline (week 1), immediately following treatment (Group 1 - week 7, Group 2 - week 13), long-term follow-up (Group 1 - week 13, Group 2 - Week 19)
  Standardized neuropsychological tests which be used will be used to determine whether there has been a change in speed of processing.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chiaravalloti, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States